CLINICAL TRIAL: NCT02942576
Title: A Prospective, Randomized, Open-Label, Blinded Endpoint Evaluation (PROBE) Parallel Group Study Comparing Edoxaban vs. VKA in Subjects Undergoing Catheter Ablation of Non-valvular Atrial Fibrillation (ELIMINATE-AF)
Brief Title: Edoxaban Treatment Versus Vitamin K Antagonist (VKA) in Patients With Atrial Fibrillation (AF) Undergoing Catheter Ablation
Acronym: ELIMINATE-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSE-EDO-01-16-EU; 2016-003069-25 (EudraCT Number)
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban; Warfarin; Phenprocoumon; fluindione; Acenocoumarol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edoxaban-based regimen (Experimental): Edoxaban-based regimen for 21 days pre- and 90 days post-ablation period.
  Interventions: Drug: Edoxaban
- VKA-based regimen (Active Comparator): VKA-based regimen for 21 days pre- and 90 days post-ablation period (control regimen)
  Interventions: Drug: VKA-Based Regimen

INTERVENTIONS:
Drug: Edoxaban — Edoxaban 60 mg once-daily or 30 mg once-daily in selected subjects.
  Other Names: Lixiana
  Arms: Edoxaban-based regimen
Drug: VKA-Based Regimen — Dosed at International Normalised Ratio (INR) levels, which is a test of how long it takes for blood to clot. Standard of Care treatment in Canada, Italy, Poland, Hungary, Czech Republic, United Kingdom (UK), Taiwan and Korea.
  Other Names: Warfarin
  Arms: VKA-based regimen
Drug: VKA-Based Regimen — Dosed at INR levels. Standard of Care treatment in Germany, Belgium, and the Netherlands.
  Other Names: Phenprogamma; Phenprocoumon
  Arms: VKA-based regimen
Drug: VKA-Based Regimen — Dosed at INR levels. Standard of Care treatment in France.
  Other Names: Previscan; Fluindione
  Arms: VKA-based regimen
Drug: VKA-Based Regimen — Dosed at INR levels. Standard of Care treatment in Spain.
  Other Names: Sintrom; Acenocoumarol
  Arms: VKA-based regimen

SUMMARY:
There are insufficient data on the safety and efficacy of edoxaban therapy in subjects with AF following catheter ablation. This phase 3b study is designed to evaluate the safety and to explore the efficacy of an edoxaban-based antithrombotic regimen versus a VKA-based antithrombotic regimen in subjects with AF following catheter ablation. Bleeding is a central safety outcome in cardiovascular clinical trials, especially for antithrombotic strategies and invasive procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age with documented history of paroxysmal (lasting ≤7 days), persistent (lasting >7 days but ≤12 months) or long-standing [long-lasting] persistent (>12 months) non-valvular AF. Duration of AF can be confirmed by any electrical tracing or a recording in the subject's medical records (e.g., medical chart, hospital discharge summary).
* Subject is eligible and is scheduled for either radio frequency (RF) or cryoballoon catheter ablation (both first and repeated procedure included).
* Signed informed consent form (ICF).

Exclusion Criteria:

* AF considered to be of a transient or reversible nature (such as in myocarditis, post-surgery, ionic disturbances, thyrotoxicosis, pneumonia, severe anemia etc.).
* Subject post stroke, or with a systemic thromboembolic event within the past 6 months prior to randomization.
* Subject has a thrombus in the left atrial appendage (LAA), left atrium (LA), left ventricle (LV), or aorta, or an intracardial mass.
* Subject had a myocardial infarction (MI) within the 2 months prior to randomization or coronary artery bypass graft (CABG) surgery within 3 months prior to the randomization.
* Subject has signs of bleeding, history of clinically-relevant bleeding according to International Society on Thrombosis and Hemostasis (ISTH), or conditions associated with high risk of bleeding
* Subjects with any contraindication for anticoagulant agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-09-24 (Actual); Study Completion 2018-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (75):
- Belgium (4):
  - ZNA Middelheim, Antwerp
  - Erasme Hospital, Brussels
  - UZ Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
- Canada (4):
  - University of Calgary, Calgary
  - Hamilton Health Sciences/McMaster University, Hamilton
  - Montreal Heart Institute, Montreal
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke
- Czechia (7):
  - FN Brno, Brno
  - St. Anne's University Hospital Brno, International Clinical Research Center, Brno
  - FN Kralovske Vinohrady, Prague
  - VFN v Praze II. Interní klinika - Kardiologie a angiologie, Prague
  - IKEM, Prague
  - University Hospital Motol - Cardiology, Prague
  - Masarykova nemocnice - Kardiologie Krajská zdravotní, a.s., Ústí nad Labem
- Germany (14):
  - Universitäts Herzzentrum Freiburg-Bad Krozingen Klinik für Kardiologie und Angiologie II, Bad Krozingen
  - Charité Universitätsmedizin Berlin - CVK Medizinische Klinik m.S. Kardiologie, Berlin
  - Klinikum Bielefeld Klinik für Kardiologie/internist. Intensivmedizin, Bielefeld
  - Klinikum Coburg GmbH II.Med.Klinik, Coburg
  - Klinik für Innere Medizin I, Dortmund
  - University Clinic Duesseldorf Clinic for Cardiology, Pneumology and Angiology, Düsseldorf
  - Universitäres Herzzentrum Hamburg Kardiologie mit Schwerpunkt Elektrophysiologie, Hamburg
  - University Hospital of Heidelberg Clinic of Cardiology, Angiology and Pneumology, Heidelberg
  - Herzzentrum Leipzig - Universitätsklinik Abteilung für Rhythmologie, Leipzig
  - Univ. of Muenster.Cardiovascular Medicine, Münster
  - Universitätsmedizin Rostock Zentrum für Innere Medizin I, Kardiologie, Rostock
  - Deutsches Herzk. Universitätsklinikum Tübingen Medizinische Klinik III. Kardiologie, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Würzburg Medizinische Klinik und Poliklinik I, Würzburg
- Hungary (6):
  - Semmelweis Egyetem Városmajori Szív- és Érgyógyászati Klinika, Budapest
  - Magyar Honvédség Egészségügyi Központ Kardiológiai Osztály, Budapest
  - Debreceni Egyetem Kardiológiai és Szívsebészeti Klinika, Debrecen
  - Pecs University Clinical Center, Pécs
  - Szegedi Tudományegyetem II. Belgyógyászati Klnika és Kardiológiai Központ, Szeged
  - Zala Megyei Szent Rafael Kórház Kardiológia Osztály, Zalaegerszeg
- Italy (14):
  - Ospedale San Donato, Arezzo
  - Pineta Grande Hospital, Castel Volturno
  - Universita' degli Studi Catanzaro, Catanzaro
  - Arcispedale Sant'Anna, Cona
  - Azienda USL Toscana, Florence
  - Ospedale della Misericordia, Grosseto
  - Ospedale dell'Angelo, Mestre
  - ASST Vimercate, Monza
  - Ospedale Santo Cuore, Negrar
  - Istituto di Cura cittè di Pavia, Pavia
  - Azienda Ospedaliera di Piacenza "Ospedale Guglielmo d Saliceto", Piacenza
  - Policlinico Casilino, Roma
  - Largo Agostino Gemelli, Rome
  - Ospedale Ecclesiastico "Miulli", Sant'Eramo
- Poland (5):
  - University Hospital - Szpital Uniwersytecki, Krakow
  - Klinika Intensywnej Terapii Kardiologicznej, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 Klinika Kardiologii, Lublin
  - Oddzial Kardiologii Szpital Grochowski im. dr R. Masztaka SPZOZ, Warsaw
  - Oddział Kliniczny Kardiologii SUM Katedra Kardiologii, Zabrze
- South Korea (5):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Yonsei University Severance Hospital, Seoul, Seodaemun-Gu
  - Korea University Anam Hospital, Seoul, Seoungbuk-gu
  - Asan Medical Center, Seoul
- Spain (5):
  - Hospital General Universitario, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Clinic Cardiologia, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario San Juan de Alicante, Sant Joan d'Alacant
- Taiwan (5):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital (VGH-TC), Taichung
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan
- United Kingdom (6):
  - Blackpool Teaching Hospitals NHS, Blackpool
  - Royal Bournemouth Hospital, Bournemouth
  - Papworth Hospital NHS Trust, Cambridge
  - Leeds General Infirmary, Leeds
  - King's College Hospital, London
  - Nottingham City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU), US and/or Japan marketing approval on or after 01 January 2014 or by the US or EU Health Authorities when regulatory submissions in both regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P, Agewall S, Camm J, Baron Esquivias G, Budts W, Carerj S, Casselman F, Coca A, De Caterina R, Deftereos S, Dobrev D, Ferro JM, Filippatos G, Fitzsimons D, Gorenek B, Guenoun M, Hohnloser SH, Kolh P, Lip GY, Manolis A, McMurray J, Ponikowski P, Rosenhek R, Ruschitzka F, Savelieva I, Sharma S, Suwalski P, Tamargo JL, Taylor CJ, Van Gelder IC, Voors AA, Windecker S, Zamorano JL, Zeppenfeld K. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Europace. 2016 Nov;18(11):1609-1678. doi: 10.1093/europace/euw295. Epub 2016 Aug 27. No abstract available. PMID 27567465
- [Background] Crawford T, Oral H. Current status and outcomes of catheter ablation for atrial fibrillation. Heart Rhythm. 2009 Dec;6(12 Suppl):S12-7. doi: 10.1016/j.hrthm.2009.07.026. Epub 2009 Oct 23. PMID 19864188
- [Background] Hussein AA, Martin DO, Saliba W, Patel D, Karim S, Batal O, Banna M, Williams-Andrews M, Sherman M, Kanj M, Bhargava M, Dresing T, Callahan T, Tchou P, Di Biase L, Beheiry S, Lindsay B, Natale A, Wazni O. Radiofrequency ablation of atrial fibrillation under therapeutic international normalized ratio: a safe and efficacious periprocedural anticoagulation strategy. Heart Rhythm. 2009 Oct;6(10):1425-9. doi: 10.1016/j.hrthm.2009.07.007. Epub 2009 Jul 10. PMID 19968920
- [Background] Cappato R, Marchlinski FE, Hohnloser SH, Naccarelli GV, Xiang J, Wilber DJ, Ma CS, Hess S, Wells DS, Juang G, Vijgen J, Hugl BJ, Balasubramaniam R, De Chillou C, Davies DW, Fields LE, Natale A; VENTURE-AF Investigators. Uninterrupted rivaroxaban vs. uninterrupted vitamin K antagonists for catheter ablation in non-valvular atrial fibrillation. Eur Heart J. 2015 Jul 21;36(28):1805-11. doi: 10.1093/eurheartj/ehv177. Epub 2015 May 14. PMID 25975659
- [Background] Chen J, Todd DM, Hocini M, Larsen TB, Bongiorni MG, Blomstrom-Lundqvist C; Scientific Initiative Committee, European Heart Rhythm Association. Current periprocedural management of ablation for atrial fibrillation in Europe: results of the European Heart Rhythm Association survey. Europace. 2014 Mar;16(3):378-81. doi: 10.1093/europace/euu043. PMID 24569891
- [Background] Hokusai-VTE Investigators; Buller HR, Decousus H, Grosso MA, Mercuri M, Middeldorp S, Prins MH, Raskob GE, Schellong SM, Schwocho L, Segers A, Shi M, Verhamme P, Wells P. Edoxaban versus warfarin for the treatment of symptomatic venous thromboembolism. N Engl J Med. 2013 Oct 10;369(15):1406-15. doi: 10.1056/NEJMoa1306638. Epub 2013 Aug 31. PMID 23991658
- [Background] Cappato R, Calkins H, Chen SA, Davies W, Iesaka Y, Kalman J, Kim YH, Klein G, Natale A, Packer D, Skanes A, Ambrogi F, Biganzoli E. Updated worldwide survey on the methods, efficacy, and safety of catheter ablation for human atrial fibrillation. Circ Arrhythm Electrophysiol. 2010 Feb;3(1):32-8. doi: 10.1161/CIRCEP.109.859116. Epub 2009 Dec 7. PMID 19995881
- [Derived] Hohnloser SH, Camm AJ, Cappato R, Diener HC, Heidbuchel H, Mont L, Morillo CA, Lanz HJ, Rauer H, Reimitz PE, Smolnik R, Kautzner J. Periprocedural anticoagulation in the uninterrupted edoxaban vs. vitamin K antagonists for ablation of atrial fibrillation (ELIMINATE-AF) trial. Europace. 2021 Jan 27;23(1):65-72. doi: 10.1093/europace/euaa199. PMID 33249467
- [Derived] Hohnloser SH, Camm J, Cappato R, Diener HC, Heidbuchel H, Lanz HJ, Mont L, Morillo CA, Smolnik R, Yin OQP, Kautzner J. Uninterrupted administration of edoxaban vs vitamin K antagonists in patients undergoing atrial fibrillation catheter ablation: Rationale and design of the ELIMINATE-AF study. Clin Cardiol. 2018 Apr;41(4):440-449. doi: 10.1002/clc.22918. Epub 2018 Apr 17. PMID 29663464

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 614 participants who met the inclusion and none of the exclusion criteria were randomized; 602 received study drug.
Pre-assignment Details: Participants were required to have completed between 21 to 28 days of anticoagulation with study treatment prior to the catheter ablation visit/periprocedural visit (Day 0).
Groups:
- VKA-based Regimen: VKA-based regimen for 21 days pre- and 90 days post-ablation period (control regimen)
  VKA-Based Regimen: Dosed at International Normalised Ratio (INR) levels, which is a test of how long it takes for blood to clot. Standard of Care treatment in Canada, Italy, Poland, Hungary, Czech Republic, UK, Taiwan and Korea.
  VKA-Based Regimen: Dosed at INR levels. Standard of Care treatment in Germany, Belgium, and the Netherlands.
  VKA-Based Regimen: Dosed at INR levels. Standard of Care treatment in France.
  VKA-Based Regimen: Dosed at INR levels. Standard of Care treatment in Spain.
Period: Overall Study
Arm/Group | Edoxaban-based Regimen | VKA-based Regimen
Started | 405 | 197
Completed | 359 | 174
Not Completed | 46 | 23
Not completed — Adverse Event | 28 | 6
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Physician Decision | 1 | 4
Not completed — Other | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- VKA-based Regimen: VKA-based regimen for 21 days pre- and 90 days post-ablation period (control regimen)
  VKA-Based Regimen: Dosed at International Normalised Ratio (INR) levels, which is a test of how long it takes for blood to clot. Standard of Care treatment in Canada, Italy, Poland, Hungary, Czech Republic, United Kingdon (UK), Taiwan and Korea.
  VKA-Based Regimen: Dosed at INR levels. Standard of Care treatment in Germany, Belgium, and the Netherlands.
  VKA-Based Regimen: Dosed at INR levels. Standard of Care treatment in France.
  VKA-Based Regimen: Dosed at INR levels. Standard of Care treatment in Spain.
- Total: Total of all reporting groups
Arm/Group | Edoxaban-based Regimen | VKA-based Regimen | Total
Number analyzed (Participants) | 405 | 197 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 262 | 130 | 392
  >=65 years | 143 | 67 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (10.2) | 59.6 (10.0) | 59.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 51 | 169
  Male | 287 | 146 | 433
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 35 | 18 | 53
  South Korea | 28 | 11 | 39
  Belgium | 5 | 4 | 9
  Hungary | 52 | 23 | 75
  Czechia | 74 | 35 | 109
  Taiwan | 25 | 14 | 39
  Poland | 54 | 24 | 78
  Italy | 42 | 21 | 63
  United Kingdom | 40 | 20 | 60
  Germany | 28 | 16 | 44
  Spain | 22 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced the Composite of All-cause Death, Stroke (VARC-2), and Major Bleeding (ISTH) in the Edoxaban Group Compared With Vitamin K Antagonist (VKA) Group in Participants Undergoing Catheter Ablation (Adjudicated Data)
Description: Stroke (ischemic, hemorrhagic, or undetermined) was defined by Valve Academic Research Consortium-2 (VARC-2) as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury following hemorrhage or infarction. A stroke event was based on any of the following: duration of neurological dysfunction >24 hours (h), duration of neurological dysfunction <24 h in case of imaging-documented new hemorrhage or infarction, and a neurological dysfunction resulting in death.
  Major bleeding was defined by the International Society on Thrombosis and Hemostasis (ISTH) as fatal bleeding and/or bleeding that is symptomatic and occurs in a critical area or organ and/or extrasurgical site bleeding causing a fall in hemoglobin level of >2 g/dL or leads to blood transfusion, surgical site bleeding that requires a second intervention, causes hemarthrosis that delays mobilization or wound healing, or causes hemodynamic instability.
Time Frame: Day 1 to Day 90
Population: The composite of all-cause death, stroke (VARC-2), and major bleeding (ISTH) was assessed in the Per Protocol (PP) Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban-based Regimen | VKA-based Regimen
Number analyzed (Participants) | 316 | 101
Participants | 1 | 2

2. Primary Outcome: Number of Participants Who Experienced Major Bleeding (International Society on Thrombosis and Hemostasis [ISTH]) in the Edoxaban Group Compared With VKA Group Among Participants Undergoing Catheter Ablation (Adjudicated Data)
Description: Major bleeding was defined by the International Society on Thrombosis and Hemostasis (ISTH) as fatal bleeding and/or bleeding that is symptomatic and occurs in a critical area or organ and/or extrasurgical site bleeding causing a fall in hemoglobin level of >2 g/dL or leads to blood transfusion, surgical site bleeding that requires a second intervention, causes hemarthrosis that delays mobilization or wound healing, or causes hemodynamic instability.
Time Frame: Day 1 to Day 90
Population: Major bleeding was assessed in the modified Intent-to-Treat (mITT) Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban-based Regimen | VKA-based Regimen
Number analyzed (Participants) | 405 | 197
Participants | 10 | 3

3. Secondary Outcome: Number of Participants Who Experienced the Composite of All-cause Death, Stroke (Alternative), and Major Bleeding (ISTH) in the Edoxaban Group Compared With VKA Group Among Participants Undergoing Catheter Ablation (Adjudicated Data)
Description: An alternative definition characterized stroke (ischemic, hemorrhagic, or undetermined) as an abrupt onset, over minutes to hours, of a focal neurological deficit in the distribution of a single brain artery that was not due to an identifiable nonvascular cause (ie, brain tumor or trauma), and that either lasted at least 24 hours or resulted in death within 24 hours of onset.
  Major bleeding was defined by the International Society on Thrombosis and Hemostasis (ISTH) as fatal bleeding and/or bleeding that is symptomatic and occurs in a critical area or organ and/or extrasurgical site bleeding causing a fall in hemoglobin level of >2 g/dL or leads to blood transfusion, surgical site bleeding that requires a second intervention, causes hemarthrosis that delays mobilization or wound healing, or causes hemodynamic instability.
Time Frame: Day 1 to Day 90
Population: The composite of all-cause death, stroke (alternative), and major bleeding (ISTH) was assessed in the PP Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban-based Regimen | VKA-based Regimen
Number analyzed (Participants) | 316 | 101
Participants | 1 | 2

4. Secondary Outcome: Number of Participants Who Experienced the Composite of Stroke (VARC-2), Systemic Embolic Events (SEE), and Cardiovascular (CV) Mortality in the Edoxaban Group Compared With VKA Group Among Participants Undergoing Catheter Ablation (Adjudicated Data)
Description: Stroke (ischemic, hemorrhagic, or undetermined) was defined by Valve Academic Research Consortium-2 (VARC-2) as an acute episode of focal or global neurological dysfunction caused by brain, spinal cord, or retinal vascular injury following hemorrhage or infarction. A stroke event was based on any of the following: duration of neurological dysfunction >24 hours (h), duration of neurological dysfunction <24 h in case of imaging-documented new hemorrhage or infarction, and a neurological dysfunction resulting in death.
  SEE was defined as an arterial embolism resulting in clinical ischemia, excluding the central nervous system, coronary, and pulmonary arterial circulation.
  CV mortality was defined as cardiac or vascular death according to Academic Research Consortium.
Time Frame: Day 1 to Day 90
Population: The composite of stroke (VARC-2), systemic embolic events (SEE), and cardiovascular (CV) mortality was assessed in the PP Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Edoxaban-based Regimen | VKA-based Regimen
Number analyzed (Participants) | 316 | 101
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the first dose of the study drug to 30 days after last dose of study drug.
Description: Adverse events that emerge (or worsen) from the first dose of the study drug to the last dose of the study drug.
Arm/Group | Edoxaban-based Regimen | VKA-based Regimen
All-Cause Mortality (participants affected / at risk) | 0/405 | 0/197
Serious Adverse Events (participants affected / at risk) | 40/405 | 15/197
Other Adverse Events (participants affected / at risk) | 210/405 | 99/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban-based Regimen (N=405) | VKA-based Regimen (N=197)
Pneumonia (Infections and infestations) | 2 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 15 | 6
Atrial flutter (Cardiac disorders) | 3 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 2
Atrial thrombosis (Cardiac disorders) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 2 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Retroperitoneal mass (Gastrointestinal disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Edoxaban-based Regimen (N=405) | VKA-based Regimen (N=197)
Atrial fibrillation (Cardiac disorders) | 41 | 21
Atrial flutter (Cardiac disorders) | 15 | 8
Palpitations (Cardiac disorders) | 12 | 4
Cardiac flutter (Cardiac disorders) | 4 | 5
Atrial tachycardia (Cardiac disorders) | 3 | 5
Pericarditis (Cardiac disorders) | 6 | 2
Nasopharyngitis (Infections and infestations) | 9 | 1
Bronchitis (Infections and infestations) | 4 | 3
Pyrexia (General disorders) | 19 | 3
Fatigue (General disorders) | 5 | 3
Non-cardiac chest pain (General disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 6 | 1
Vomiting (Gastrointestinal disorders) | 5 | 2
Abdominal pain upper (Gastrointestinal disorders) | 5 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 3
Headache (Nervous system disorders) | 8 | 5
Dizziness (Nervous system disorders) | 8 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Alanine aminotransferase increased (Investigations) | 5 | 0
Hypertension (Vascular disorders) | 8 | 3
Hypotension (Vascular disorders) | 8 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Hypokalemia (Metabolism and nutrition disorders) | 2 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 | 2
Phrenic nerve paralysis (Nervous system disorders) | 1 | 2
Atrioventricular block first degree (Cardiac disorders) | 3 | 2
Atrial thrombosis (Cardiac disorders) | 2 | 2
Bradycardia (Cardiac disorders) | 0 | 2
Arteriovenous fistula (Vascular disorders) | 3 | 2
Flatulence (Gastrointestinal disorders) | 2 | 2
Liver disorder (Hepatobiliary disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Renal impairment (Renal and urinary disorders) | 2 | 2
Procedural pain (Injury, poisoning and procedural complications) | 4 | 2
Post procedural complication (Injury, poisoning and procedural complications) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT02942576/Prot_SAP_000.pdf